CLINICAL TRIAL: NCT01810003
Title: Impact of EPA and DHA Supplementation on Plasma Biomarkers of Inflammation in Men and Women With Metabolic Syndrome
Brief Title: Impact of EPA and DHA Supplementation on Plasma Biomarkers of Inflammation (n3)
Acronym: n3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-2012-143
Record Dates: First submitted 2013-03-04; First posted 2013-03-13 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Disease, Inflammation
Keywords: Cardiovascular disease; Inflammation; EPA/DHA supplementation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High DHA (Experimental): High DHA supplementation (3g/day)
  Interventions: Dietary Supplement: High DHA
- High EPA (Experimental): EPA supplementation (3g/day)
  Interventions: Dietary Supplement: High EPA
- Placebo (Placebo Comparator): Placebo (3g corn oil/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High DHA — 10 week supplementation period
  Arms: High DHA
Dietary Supplement: High EPA — 10 week supplementation period
  Arms: High EPA
Dietary Supplement: Placebo — 10 week supplementation period
  Arms: Placebo

SUMMARY:
Subclinical inflammation is now indisputably recognized as a key etiological factor in the development of atherosclerosis and subsequent cardiovascular disease. Obesity and related dysmetabolic states including metabolic syndrome (MetS) are highly prevalent causes of subclinical inflammation. Obesity and MetS are both diet and lifestyle-related and there is a growing body of literature suggesting that specific nutrients, such as long chain omega-3 polyunsaturated fatty acids (LCn-3PUFA), may attenuate the pro-inflammatory state associated with these conditions. However, careful review of existing literature on this topic reveals important gaps in knowledge, the purported anti-inflammatory effects of LCn-3PUFA even being questioned by many. Significant confounding attributable to study design, sample size and biomarker selection may be responsible in part for inconsistencies in the literature on LCn-3PUFA and inflammation. We also found that evidence available to date (for and against) is based primarily on secondary analyses, as most of the studies published were not primarily designed to investigate inflammation as a primary outcome. It remains unclear whether the different LCn-3PUFA, primarily docosahexaenoic acid (DHA, 22:6n-3) and eicosapentaenoic acid (EPA, 20:5n-3), have similar effects on pro-inflammatory processes as almost all studies were undertaken using a mix of LCn-3PUFA. Whether efficacy of EPA and DHA is influenced by sex/gender is also unknown. Finally, a better understanding of the systemic and tissue-specific mechanisms underlying the anticipated anti-inflammatory effects of different LCn-3PUFA in MetS would also be of great value. Addressing these gaps has important public health implications, considering that LCn-3PUFA supplements are broadly and indiscriminately recommended for the prevention of cardiovascular disease.

The overarching objective of the proposed research is to compare the anti-inflammatory effects of EPA and DHA in men and women with MetS.

DETAILED DESCRIPTION:
The proposed study will be undertaken according to a double-blind randomized placebo controlled cross-over design with 3 treatment phases: 1- high DHA, 2- High EPA, 3- Control. Each treatment phase will last 10 weeks and will be separated by 8-week washouts. Participants will be randomized to one of 6 treatment sequences while stratifying for sex. Treatments will provide 3 identical 1g capsules per day. During the 3 treatment periods, subjects will receive in random order 0g/d EPA+DHA (3g corn oil placebo), 3g/d EPA (>90% EPA), and 3g/d DHA (>90% DHA). Long chain omega-3 polyunsaturated fatty acids (LCn-3PUFA) will be provided in their re-esterified triacylglycerol form as studies have shown that bioavailability was greater when EPA and DHA were consumed as TG rather than as ethyl esters. The therapeutic dose that maximizes the anti-inflammatory effects of LCn-3PUFA in patients with inflammation has not been established, although data suggest that they may be dose-dependent. However, studies in healthy human volunteers suggest that an intake > 2 g EPA + DHA/day is required to affect inflammatory processes. Many of the available studies have used a dose of EPA+DHA that was lower than 2g/d, with no apparent anti-inflammatory effects. A study has shown that a dose of 1.8g/d of EPA+DHA induced significant changes in peripheral blood cell (PBC) inflammation gene expression, with no change in plasma CRP concentrations. In the present study, we propose to use a dose of 3 g/d for each individual LCn-3PUFA tested, which is at the higher end of the recommended intake for patients with high plasma TG, but which will maximize our chance to observe changes in inflammatory markers and to differentiate the effects of EPA and DHA, if they exist. Participants will be instructed to maintain a constant body weight during the course of the study. They will also be counselled on how to exclude fatty fish meals (including salmon, tuna, mackerel, and herring), fish-oil supplements, flax products, walnuts, and omega-3-enriched eggs during the study. Vitamin supplements and natural health products will be strictly forbidden during the entire experimental period, with the exception of calcium and vitamin D, which will be allowed at a stable dose. Although alcohol consumption will be permitted during the study with intakes not exceeding one serving (12-15 g alcohol) per day, it will be forbidden for the 4 days that precede the various tests at the end of each treatment phase. Subjects will also be instructed to maintain their usual physical activity except for the 4 days that precede blood sampling at the various stages of the study, during which they will be asked to remain sedentary.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years with abdominal obesity as defined by the International Diabetes Federation criteria and a measure of plasma CRP >1 mg/L
* Stable body weight for at least 3 months prior to randomization.
* Pre-menopausal women with regular menstrual cycle (25-35 days)

Exclusion Criteria:

* Plasma CRP > 10 mg/L at screening
* Extreme dyslipidemias such as familial hypercholesterolemia
* Previous history of cardiovascular disease (coronary heart disease, cerebrovascular disease or peripheral arterial disease)
* Subjects taking medications known to affect inflammation (e.g. steroids, binging alcohol)
* Subjects taking LCn-3PUFA supplements within 2 months of study onset.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma biomarkers of inflammation (CRP, Interleukin (IL)-6, IL-18 and Tumor necrosis factor-α) | At the beginning and the end of each 10-week period
  Change between treatments based on post-treatment values, adjusting for treatment-specific baseline values

SECONDARY OUTCOMES:
Change in lipid concentrations (LDL-C, HDL-C, TG) | At the beginning and the end of each 10-week period
  Change between treatments based on post-treatment values, adjusting for treatment-specific baseline values
Change in blood pressure | At the beginning and the end of each 10-week period
  Change between treatments based on post-treatment values, adjusting for treatment-specific baseline values
Change in endogenous production and clearance rate of CRP (in a subsample of the entire study population) | At the end of the three 10-week periods
  Change between treatments based on post-treatment values
Change in expression of inflammation genes in peripheral blood cells (in a subsample of the entire study population) | At the end of the three 10-week periods
  Change between treatments based on post-treatment values
Change in anthropometric measures (waist and hip circumference) | At the beginning and the end of each 10-week period
  Change between treatments based on post-treatment values, adjusting for treatment-specific baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Vallee Marcotte B, Allaire J, Guenard F, de Toro-Martin J, Couture P, Lamarche B, Vohl MC. Genetic risk prediction of the plasma triglyceride response to independent supplementations with eicosapentaenoic and docosahexaenoic acids: the ComparED Study. Genes Nutr. 2020 Jun 15;15(1):10. doi: 10.1186/s12263-020-00669-x. PMID 32539794
- [Derived] Allaire J, Vors C, Tremblay AJ, Marin J, Charest A, Tchernof A, Couture P, Lamarche B. High-Dose DHA Has More Profound Effects on LDL-Related Features Than High-Dose EPA: The ComparED Study. J Clin Endocrinol Metab. 2018 Aug 1;103(8):2909-2917. doi: 10.1210/jc.2017-02745. PMID 29846653
- [Derived] Vors C, Allaire J, Marin J, Lepine MC, Charest A, Tchernof A, Couture P, Lamarche B. Inflammatory gene expression in whole blood cells after EPA vs. DHA supplementation: Results from the ComparED study. Atherosclerosis. 2017 Feb;257:116-122. doi: 10.1016/j.atherosclerosis.2017.01.025. Epub 2017 Jan 20. PMID 28131045
- [Derived] Allaire J, Couture P, Leclerc M, Charest A, Marin J, Lepine MC, Talbot D, Tchernof A, Lamarche B. A randomized, crossover, head-to-head comparison of eicosapentaenoic acid and docosahexaenoic acid supplementation to reduce inflammation markers in men and women: the Comparing EPA to DHA (ComparED) Study. Am J Clin Nutr. 2016 Aug;104(2):280-7. doi: 10.3945/ajcn.116.131896. Epub 2016 Jun 8. PMID 27281302